CLINICAL TRIAL: NCT06658405
Title: Phase 2 Clinical Trial Evaluating Secondary HPV Vaccination After Treatment of High-grade Cervical Lesions (HPV2-2303)
Brief Title: Clinical Trial Evaluating Secondary HPV Vaccination After Treatment of High-grade Cervical Lesions
Acronym: HPV2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPV2-2303; 2024-513081-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-02

CONDITIONS: Cervical Lesion
Keywords: HPV; oncology; secondary prevention; cervix; vaccination
MeSH Terms: conditions — Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Intervention Model Description: The study uses a non-randomized design with two cohorts: vaccinated patients in a single-arm clinical trial and non-vaccinated patients in an observational study, chosen to reflect real-life scenarios and ensure comprehensive data collection despite the absence of randomization..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccinated patients (Experimental): Human papillomavirus vaccine, nonvalent, Gardasil 9
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant
- Non-vaccinated patients (No Intervention): no changes to standard care

INTERVENTIONS:
Biological: Human Papillomavirus 9-valent Vaccine, Recombinant — HPV vaccine administered in three doses: first dose on day 1, second dose 2 months later, and third dose 4 months after the second dose, within a one-year period.
  Other Names: Gardasil 9
  Arms: Vaccinated patients

SUMMARY:
This is a single-center, Phase II interventional study evaluating secondary HPV vaccination after treatment of high-grade cervical lesions. The study aims to estimate the rate of HPV clearance within two years following an initial positive HPV control test in women over 45 years of age who are chronic HPV carriers and have undergone treatment for high-grade intraepithelial cervical lesions, and who receive HPV vaccination.

The study includes two cohorts:

1. Eligible patients who consent to vaccination will participate in a prospective, single-center, single-arm, interventional clinical trial (Category 2).
2. Non-vaccinated patients will be included in a non-interventional observational study, with no changes to their standard care.

DETAILED DESCRIPTION:
The aim of this study is to estimate the proportion of HPV clearance within two years following an initial positive HPV control test in women over 45 years old who are chronic HPV carriers and have undergone treatment for high-grade intraepithelial cervical lesions. These women will receive HPV vaccination as part of the study.

Other objectives of the study include:

1. Describing the dynamics of viral clearance in chronic HPV carriers who receive HPV vaccination.
2. Evaluating the safety of HPV vaccination.
3. Estimating the incidence of recurrence of high-grade intraepithelial cervical lesions in chronic HPV carriers after surgical treatment of the initial lesion and HPV vaccination.
4. Estimating the incidence of invasive gynecological cancers (cervical, vaginal, or vulvar) in chronic HPV carriers after surgical treatment of the initial lesion and HPV vaccination.
5. Identifying factors associated with the refusal of HPV vaccination, such as smoking, parity, body mass index, employment status, education level, family history, and marital status.
6. Describing compliance with the proposed vaccination schedule in terms of:

   1. Number of injections completed.
   2. Adherence to the timing of injections.
7. Evaluating the effect of vaccination on:

   1. HPV clearance within two years.
   2. The dynamics of viral clearance.
   3. The risk of recurrence of high-grade intraepithelial lesions.
   4. The risk of developing invasive gynecological cancers (cervical, vaginal, or vulvar).

by comparing vaccinated patients included in the clinical trial with the cohort of non-vaccinated patients (those who refused HPV vaccination or for other reasons).

ELIGIBILITY:
Inclusion Criteria:

1. Common eligibility criteria for the study (for both cohorts) :

   1. Female patient over 45 years old
   2. Patient treated by conization for high-grade cervical epithelial lesion
   3. Positive HPV test at the 6-month post-operative control (a delay of 6 to 12 months will be accepted), leading to an indication for a control colposcopy (+/- biopsy) according to standard surveillance practices.
   4. N.B. : Patients with abnormalities at the initial control colposcopy and/or positive biopsy remain eligible for the study, whether vaccinated or not.
2. Additional eligibility criteria for the clinical trial (Vaccinated patients cohort)

   1. No contraindication to HPV vaccination with Gardasil 9
   2. Patient consented to HPV vaccination with Gardasil 9
   3. Affiliated with a social security system
   4. Informed and signed written consent provided
   5. N.B. : Patients infected with HIV are eligible for the vaccine trial provided they are on antiretroviral therapy.
3. Inclusion criteria for the data study (Non-vaccinated patients cohort)

   1. Patient eligible for the study (a) and not eligible for the clinical trial (b) due to:

      * refusal of vaccination, or
      * A contraindication to vaccination
   2. No objection to the use of their personal data for research purposes

N.B. : A patient who initially refused vaccination may later request to be vaccinated as part of the trial after signing the consent form. The vaccine trial analysis will include all patients who started vaccination within 6 months after the initial HPV control test.

Exclusion Criteria:

1. Common exclusion criteria for the study (for both cohorts)

   1. History of primary HPV vaccination
   2. History of HPV-induced invasive cancer (cervical, vaginal, vulvar, anal, oropharyngeal cancer)
2. Exclusion criteria for the clinical trial (Vaccinated patients cohort)

   1. Patient refusing HPV vaccination
   2. Patient with a contraindication to HPV vaccination with Gardasil 9
   3. Patient deprived of liberty or under guardianship
3. Exclusion criteria for the data study (Non-vaccinated patients cohort) a) Opposition to the use of their personal data for research purposes

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with chronic HPV infections, particularly those who have undergone treatment for high-grade cervical lesions.
Enrollment: 85 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of HPV-negative status | Within 2 years after the initial HPV control test
  The primary outcome is to estimate the proportion of HPV-negativation status within two years of the initial positive HPV control test. Negativation is defined as a negative HPV test result. If the patient cannot be evaluated due to the occurrence of cancer, this will be considered a failure (equivalent to absence of negativation).

SECONDARY OUTCOMES:
Dynamics of HPV viral clearance | every 12 months for up to 5 years
  HPV status over time assessed by smear every 12 months until HPV-negative status (in the study: within 5 years of follow-up). When the test is negative, a follow-up smear is performed three years later (in the study: within 5 years of follow-up)
Adverse Events | Throughout the vaccination schedule plus 30 days
  Adverse events will be recorded and evaluated according to the NCI-CTCAE V5.0 scale. AEs will be documented after each vaccination, during subsequent injections, and through a follow-up phone call 30 days after the third injection. Severe Adverse Events (grade ≥3) will be considered significant.
Incidence of high-grade intraepithelial lesions | From the initial HPV control test up to the first recurrence event up to 5 years
  The time to recurrence of high-grade cervical lesions will be calculated from the date of the initial HPV control test to the first documented event of lesion recurrence, as indicated by clinical follow-up and diagnostic testing.
Incidence of invasive gynecological cancer | From the initial HPV control test to the occurrence of invasive cancer up to 5 years
  The incidence of invasive gynecological cancers (cervix, vagina, vulva) will be determined by calculating the time from the initial HPV control test to the first occurrence of HPV-related invasive cancer at any sites (cervix, vagina, vulva)
Compliance with vaccination schedule | Throughout the vaccination period (up to 1 year)
  Compliance will be measured by the number of vaccine doses received and adherence to the recommended timing between injections, including the interval between the 1st and 3rd doses of Gardasil 9.

CONTACTS AND LOCATIONS:
Overall Officials: Nora ALLOY, MD, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No